CLINICAL TRIAL: NCT07261969
Title: CRP and Patient Information Leaflets to Optimise Antibiotic Treatments for Adults With Respiratory Tract Infections in Primary Care in Kyrgyzstan
Acronym: 2CARE INSTALL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: International Centre for Antimicrobial Resistance Solutions (ICARS) (Unknown); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jesper Kjærgaard, Head of the unit for children and adolescents with infections or organ-disease, Rigshospitalet, Denmark
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: INSTALL WP1
Record Dates: First submitted 2024-12-18; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2024-12

CONDITIONS: Respiratory Tract Infection Bacterial; Respiratory Tract Infection Viral; AMR; CRP; Inflammation
Keywords: CRP POCT; Primary care; ARVI; ARTI; Adults; PIL; RCT
MeSH Terms: conditions — Inflammation | interventions — World Health Organization

STUDY DESIGN:
Intervention Model Description: A multicentre, open-label, individually randomised controlled clinical trial with 21 days blinded follow-up comparing PIL to no PIL in a 1:1 ratio on antibiotic use and safety. Additionally, antibiotic use and safety will be assessed across three CRP cut-offs (20-40-60 mg/L) in a 1:1:1 ratio to determine the optimal CRP cut-offs in these cohorts. Thus, in total, six groups will be randomly formed and compared. The trial will be conducted in 14 selected district primary-level Healthcare Centres (HCs) in rural Kyrgyzstan and one urban primary-level HC in Bishkek.
Who Masked: Outcomes Assessor
Masking Description: Following the baseline consultation, follow-up calls will be made to the telephone number provided by the participants on days 3, 7, 14 and 21 (Figure 1) by a blinded researcher from the Bishkek office.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group AX (Active Comparator): This arm will receive the CRP POCT intervention plus patient information leaflet. The threshold values of CRP for this group are 20 mg/l.
  Interventions: Diagnostic Test: The C-reactive protein point-of-care test (CRP-POCT); Behavioral: Patient information leaflets
- Group AY (Active Comparator): This arm will receive the CRP POCT intervention plus patient information leaflet. The threshold values of CRP for this group are 40 mg/l.
  Interventions: Diagnostic Test: The C-reactive protein point-of-care test (CRP-POCT); Behavioral: Patient information leaflets
- Group AZ (Active Comparator): This arm will receive the CRP POCT intervention plus patient information leaflet. The threshold values of CRP for this group are 60 mg/l.
  Interventions: Diagnostic Test: The C-reactive protein point-of-care test (CRP-POCT); Behavioral: Patient information leaflets
- Group BX (Active Comparator): This arm will receive only the CRP POCT intervention. The threshold values of CRP for this group are 20 mg/l.
  Interventions: Diagnostic Test: The C-reactive protein point-of-care test (CRP-POCT)
- Group BY (Active Comparator): This arm will receive only the CRP POCT intervention. The threshold values of CRP for this group are 40 mg/l.
  Interventions: Diagnostic Test: The C-reactive protein point-of-care test (CRP-POCT)
- Group BZ (Active Comparator): This arm will receive only the CRP POCT intervention. The threshold values of CRP for this group are 60 mg/l.
  Interventions: Diagnostic Test: The C-reactive protein point-of-care test (CRP-POCT)

INTERVENTIONS:
Diagnostic Test: The C-reactive protein point-of-care test (CRP-POCT) — The intervention involves using the Aidian QuickRead go system, a portable, user-friendly device designed for point-of-care testing. This system provides rapid and reliable results for various tests, including C-reactive protein (CRP) levels, which help in diagnosing and managing infections. The device features an intuitive touch screen, minimal hands-on time, and secure data storage, making it an effective tool for guiding antibiotic use in primary healthcare settings.
  Other Names: Aidian QuickRead go (Espoo, Finland)
Behavioral: Patient information leaflets — The WHO's antibiotic-free prescription intervention aims to reduce unnecessary antibiotic use by providing clear guidelines and educational materials to healthcare providers and patients. This intervention includes Patient Information Leaflet (PIL) that explain when antibiotics are not needed, such as for viral infections, and promote alternative symptom management strategies (symptomatic).
  Other Names: Antiobiotic-free prescription produced by WHO
  Arms: Group AX; Group AY; Group AZ

SUMMARY:
This study aims to determine how CRP levels and Patient Information Leaflets (PILs) affect antibiotic prescribing in adults with acute respiratory symptoms in Kyrgyz primary care. It will evaluate the effectiveness of PILs in reducing antibiotic use and ensuring safety and assess the effectiveness and safety of three CRP thresholds (20, 40, 60 mg/L) for adults with acute respiratory tract infections. Conducted as a multicentre, open label, individually randomized controlled clinical trial with 21 days of blinded follow-up, the study will compare PIL to no PIL in a 1:1 ratio and assess antibiotic use and safety across the three CRP cut-offs in a 1:1:1 ratio, resulting in six groups. The trial will take place in 14 district primary healthcare centres in rural Kyrgyzstan and one urban primary healthcare centre in Bishkek.

DETAILED DESCRIPTION:
BACKGROUND Antimicrobial resistance (AMR) poses a significant global health threat, particularly in Kyrgyzstan, where overuse and misuse of antibiotics have fueled the crisis. The easy over-the-counter availability of antibiotics has led to widespread misuse, escalating resistance among common pathogens. This undermines effective treatment for infections, increasing healthcare costs and mortality rates. Although Kyrgyzstan is part of the Central Asian and European Surveillance of Antimicrobial Resistance (CAESAR) network, it faces challenges such as inadequate data reporting, limited resources, and insufficient training in rational antibiotic use. Efforts are underway, including a national action plan and a CIS-wide joint initiative to address AMR, focusing on public education, vaccination, and healthcare training. Improved diagnostic tools like C-reactive protein (CRP) testing have shown promise in reducing unnecessary antibiotic prescriptions by distinguishing between bacterial and viral infections.

The COORDINATE trial in Kyrgyzstan demonstrated that CRP point-of-care testing (POCT) effectively reduces antibiotic use for respiratory tract infections (RTIs) without compromising patient safety. The study's findings prompted the Ministry of Health to plan nationwide implementation of CRP POCT in primary healthcare. However, further research is needed to establish appropriate CRP thresholds for adults. Complementary strategies such as antibiotic-free patient information leaflets (PILs) can educate the public on appropriate antibiotic use, promoting alternative symptom management and reducing patient demand for unnecessary prescriptions. Together, these measures can improve antibiotic stewardship, mitigate AMR, and enhance public health outcomes.

The research team will address these challenges in the 2CARE study:

1. an adequate understanding of the AMR context may work together with the use of CRP POCT to additionally lower antibiotic use. Hence, this understanding needs to be instilled in the patient. To aid in this, the use of written materials (PILs) in the consultation is evaluated in the present study.
2. What CRP-threshold to choose: a low threshold may not lower antibiotic use much, while a high threshold could significantly reduce antibiotic use, but possibly at the expense of a higher rate of adverse events (hospitalisations, longer recovery times) due to the risk of undertreatment of bacterial pneumonia. In order to identify relevant thresholds, guidelines are reviewed to assess which CRP values are applied in adult patients who present with acute respiratory infection.

AIM The study aims to determine how CRP levels and PILs affects antibiotic prescribing in adults presenting with acute respiratory symptoms in Kyrgyz primary care.

OBJECTIVES

1. To evaluate the effectiveness of PILs to reduce the participants' tendency to take antibiotics and the safety of PILs with respect to not increase hospitalisations.
2. To evaluate the effectiveness and safety of selected CRP thresholds (low, middle, high) for adults with acute respiratory tract infection.

STUDY SETTING The study will integrate healthcare centres (HCs) from the COORDINATE trial and newly selected sites, chosen based on logistical convenience, transport infrastructure, and patient flow. Primary healthcare workers (HCWs), including family doctors, nurses, and feldshers in rural clinics with limited equipment, will participate. HCWs from new sites will receive training in CRP testing, interpretation, and providing patient information leaflets (PILs), while those from COORDINATE sites will refresh their skills. Training will use the Aidian QuickRead Go device and cover CRP threshold values. Site-specific characteristics will be addressed in covariate analysis and subgroup analysis to understand their impact on healthcare delivery and outcomes.

PARTICIPANTS Adult patients aged 18 to 70 years with acute respiratory tract infections (ARTIs) and symptoms such as cough, shortness of breath, sore throat, stuffy nose, or wheezing lasting less than two weeks will be screened during normal working hours over two winter and early spring periods (2025 and 2026) at 15 selected primary healthcare centres. Eligible participants must provide written informed consent and comply with study requirements. Exclusion criteria include severe or terminal illness, immunosuppression, recent antibiotic use, pregnancy, inability to participate in follow-up, or unwillingness to provide consent.

PROCEDURES The research team will screen patients at healthcare centres to identify eligible participants, who will provide informed consent in written or oral form. Patients of any ethnicity and both sexes, aged up to 70 years, will be included due to the average life expectancy in Kyrgyzstan. Upon enrollment, the research team will contact an investigator at the central office in Bishkek to assign a unique participant ID and randomise the participant into one of six groups. All subsequent study procedures will take place in the healthcare worker's office, typically involving a physician or feldsher, often assisted by a nurse.

INTERVENTION All participants will undergo CRP POCT testing during their consultation with a pre-trained healthcare worker (HCW) using the Aidian QuickRead Go device. Antibiotic prescriptions will follow the assigned CRP cut-off subgroup (>20 mg/L, >40 mg/L, >60 mg/L), with results recorded in the case report form (CRF) and explained to patients in plain language. In Groups A (AX, AY, AZ), participants will also receive a patient information leaflet (PIL), regardless of antibiotic prescription, emphasizing the importance of avoiding antibiotics for low CRP levels when a viral infection is suspected. Follow-up calls will be conducted by blinded researchers on days 3, 7, 14, and 21, and all participants will be advised to seek further care if symptoms worsen or fail to improve, following standard ARTI management practices in Kyrgyzstan.

CRITERIA FOR DISCONDUCTING FOR MODIGYING INTERVENTIONS Each participant will be involved in the trial for 21 days to report any adverse events (AEs), with serious adverse events (SAEs) reviewed by a safety board comprising the primary investigator, a biostatistician, and three academic members (one Kyrgyz and two Danish). SAEs must be reported to the primary investigator within 24 hours and to the safety board within 14 days. The safety board can terminate the trial if safety concerns arise, and participants will be informed and provided follow-up care if the trial ends prematurely. Discontinuation from the trial may occur due to withdrawn consent or protocol violations, but participants are not required to provide reasons. AEs leading to discontinuation will be followed up, and data collected until discontinuation will be included in the analysis. Exclusion criteria met during the follow-up period will not automatically result in discontinuation, and participants will not be replaced.

SAMPLE SIZE AND POWER CALCULATION The study aims to recruit 1,050 participants to evaluate both primary outcomes while accounting for up to 5% loss to follow-up. To detect a 10 percentage point reduction in antibiotic use with patient information leaflets (PILs) (from 40% to 30%) with 90% power and 5% significance, 1,012 participants are required. For the safety outcome, ensuring non-inferiority with a 5 percentage point margin in hospitalisation rates (expected at 5%) requires 978 participants. These calculations ensure adequate power to assess the study's primary outcomes reliably.

STATISTICAL METHODS The study will analyze baseline characteristics, such as living place, age, sex, and occupation, using medians with interquartile ranges for continuous variables (tested with the Kruskal-Wallis test) and percentages for categorical variables (tested with chi-squared tests). Outcomes will be assessed as risk differences (RD) through linear regression and odds ratios (OR) via logistic regression, with adjustments for correlations using Generalized Estimating Equations (GEE). The effects of the PIL and CRP interventions will be analyzed separately, with adjustments for the other intervention. An interim analysis will be conducted after 500 participants (50% of the target), allowing for early trial termination if interventions show clear benefits, harm, or futility. Subgroup analyses will explore outcomes by age group (18-44/45-59/60-70), urban/rural settings, clinic type, and sex.

TRIAL STATUS Protocol version 2.1. December 2nd, 2024. Date of start recruitment estimated to be January 2025. Estimated end of recruitment March 2026

DECLARATIONS Ethics approval and consent to participate Ethical approval for the 2CARE RCT was obtained during a meeting of the Ethics Committee, which included the chairman and other members of the Ethics Committee of the National Centre of Cardiology and Internal Medicine named after academician M. Mirrakhimov. During the meeting, the study protocol was reviewed, and the principal investigator addressed questions regarding the intervention. The decision was documented and signed by each member (Ref. No 10 27.11.2024). As stated earlier, before inclusion in the study, the participant will be asked to sign an informed consent, otherwise the participant cannot be included in the study. The informed consent is on the first page of the CRF.

COMPETING INTERESTS There are no competing interests.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 70 years with ARTI according to the attending HCW;
* Having at least one of the following respiratory symptoms lasting for less than 2 weeks (with or without a fever):

  * cough;
  * shortness of breath;
  * sore throat;
  * stuffy nose;
  * wheezing.
* Able and willing to comply with all study requirements.
* Able and willing to give informed consent.

Exclusion Criteria:

* Severely ill and in need of urgent referral where measurement of POCT CRP is not relevant or would delay the process;
* Terminally ill patients;
* Patients with known immunosuppression or severe chronic disease (HIV, liver failure, kidney failure, history of neoplastic disease, long term systemic steroid use or similar conditions as assessed by the health worker or research team);
* Patients who are not able to participate in follow-up procedures (lack of telephone etc.);
* Have taken antibiotics within 24 hours before the index consultation;
* Pregnant women;
* Unable or unwilling to provide informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome (mainly relevant relative to the PIL intervention) | Over 21 days.
  The rate of total antibiotic prescriptions (prescribed as well as non-prescribed (e.g. purchased over the counter or taken from home storage).
The second primary outcome (mainly relevant relative to the CRP threshold intervention) | Over 21 days.
  The safety measured as a rate of hospital admissions.

SECONDARY OUTCOMES:
Secondary study outcomes | At baseline assessment (Day 0) and over 21 days.
  The rate of antibiotic prescriptions at the baseline assessment; self-reported recovery (rate of responses from participants indicating their recovery; mortality (rate of deaths); rate of antibiotic use started outside of health care visits; rate of antiviral treatment prescriptions; rate of re-consultations; rate of hospital referral at the baseline consultation.

CONTACTS AND LOCATIONS:
Locations (2):
- Kyrgyzstan (2):
  - Sokuluk Family Medicine Center, Sokuluk Village, Chui Region
  - Azim Azhybek uulu, At-Bashy Village, Naryn Region

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data (IPDs).

REFERENCES:
- [Background] Antimicrobial Resistance Collaborators. Global burden of bacterial antimicrobial resistance in 2019: a systematic analysis. Lancet. 2022 Feb 12;399(10325):629-655. doi: 10.1016/S0140-6736(21)02724-0. Epub 2022 Jan 19. PMID 35065702
- [Background] Holmes AH, Moore LS, Sundsfjord A, Steinbakk M, Regmi S, Karkey A, Guerin PJ, Piddock LJ. Understanding the mechanisms and drivers of antimicrobial resistance. Lancet. 2016 Jan 9;387(10014):176-87. doi: 10.1016/S0140-6736(15)00473-0. Epub 2015 Nov 18. PMID 26603922
- [Background] Munita JM, Arias CA. Mechanisms of Antibiotic Resistance. Microbiol Spectr. 2016 Apr;4(2):10.1128/microbiolspec.VMBF-0016-2015. doi: 10.1128/microbiolspec.VMBF-0016-2015. PMID 27227291
- [Background] Baktygul K, Marat B, Ashirali Z, Harun-Or-rashid M, Sakamoto J. An assessment of antibiotics prescribed at the secondary health-care level in the Kyrgyz Republic. Nagoya J Med Sci. 2011 Aug;73(3-4):157-68. PMID 21928697
- [Background] Do NTT, Vu TVD, Greer RC, Dittrich S, Vandendorpe M, Pham NT, Ta DN, Cao HT, Khuong TV, Le TBT, Duong TH, Nguyen TH, Cai NTH, Nguyen TQT, Trinh ST, van Doorn HR, Lubell Y, Lewycka S. Implementation of point-of-care testing of C-reactive protein concentrations to improve antibiotic targeting in respiratory illness in Vietnamese primary care: a pragmatic cluster-randomised controlled trial. Lancet Infect Dis. 2023 Sep;23(9):1085-1094. doi: 10.1016/S1473-3099(23)00125-1. Epub 2023 May 22. PMID 37230105
- [Background] Smedemark SA, Aabenhus R, Llor C, Fournaise A, Olsen O, Jorgensen KJ. Biomarkers as point-of-care tests to guide prescription of antibiotics in people with acute respiratory infections in primary care. Cochrane Database Syst Rev. 2022 Oct 17;10(10):CD010130. doi: 10.1002/14651858.CD010130.pub3. PMID 36250577
- [Background] Isaeva E, Bloch J, Poulsen A, Kurtzhals J, Reventlow S, Siersma V, Akylbekov A, Sooronbaev T, Munck Aabenhus R, Kjaergaard J. C reactive protein-guided prescription of antibiotics for children under 12 years with respiratory symptoms in Kyrgyzstan: protocol for a randomised controlled clinical trial with 14 days follow-up. BMJ Open. 2023 Apr 11;13(4):e066806. doi: 10.1136/bmjopen-2022-066806. PMID 37041063
- [Background] Ngwengi Y, Ngaba GP, Nida M, Enyama D. Evaluation of CRP as a marker for bacterial infection and malaria in febrile children at the Douala Gyneco-Obstetric and Pediatric Hospital. PLoS One. 2023 Jul 21;18(7):e0289012. doi: 10.1371/journal.pone.0289012. eCollection 2023. PMID 37478118
- [Background] Escadafal C, Incardona S, Fernandez-Carballo BL, Dittrich S. The good and the bad: using C reactive protein to distinguish bacterial from non-bacterial infection among febrile patients in low-resource settings. BMJ Glob Health. 2020 May;5(5):e002396. doi: 10.1136/bmjgh-2020-002396. PMID 32467355
- [Background] Sustersic M, Gauchet A, Foote A, Bosson JL. How best to use and evaluate Patient Information Leaflets given during a consultation: a systematic review of literature reviews. Health Expect. 2017 Aug;20(4):531-542. doi: 10.1111/hex.12487. Epub 2016 Sep 26. PMID 27669682
- [Background] de Bont EG, Alink M, Falkenberg FC, Dinant GJ, Cals JW. Patient information leaflets to reduce antibiotic use and reconsultation rates in general practice: a systematic review. BMJ Open. 2015 Jun 3;5(6):e007612. doi: 10.1136/bmjopen-2015-007612. PMID 26041493
- [Background] Wyczalkowska-Tomasik A, Czarkowska-Paczek B, Zielenkiewicz M, Paczek L. Inflammatory Markers Change with Age, but do not Fall Beyond Reported Normal Ranges. Arch Immunol Ther Exp (Warsz). 2016 Jun;64(3):249-54. doi: 10.1007/s00005-015-0357-7. Epub 2015 Aug 18. PMID 26283530
- [Background] Williamson SF, Grayling MJ, Mander AP, Noor NM, Savage JS, Yap C, Wason JMS. Subgroup analyses in randomized controlled trials frequently categorized continuous subgroup information. J Clin Epidemiol. 2022 Oct;150:72-79. doi: 10.1016/j.jclinepi.2022.06.017. Epub 2022 Jul 2. PMID 35788399
- See also: O'Neill J. Tackling drug-resistant infections globally: Final report and recommendations. Review on Antimicrobial Resistance. 2016. — https://amr-review.org/sites/default/files/160518_Final%20paper_with%20cover.pdf
- See also: Central Asian and European Surveillance of Antimicrobial Resistance Annual Report 2020. — https://iris.who.int/handle/10665/345873
- See also: Global antimicrobial resistance and use surveillance system (GLASS) report: 2022 — https://www.who.int/publications/i/item/9789240062702
- See also: Influenza and ARVI in Kyrgyzstan — https://iimmun.ru/iimm/article/view/248
- See also: Life expectancy at birth, total (years) - Kyrgyz Republic — https://data.worldbank.org/indicator/SP.DYN.LE00.IN?locations=KG
- See also: QuikRead go Instrument — https://www.aidian.eu/point-of-care/quikread-go/quikread-go-instrument

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT07261969/Prot_SAP_000.pdf